CLINICAL TRIAL: NCT05707182
Title: 18F-rhPSMA-7.3 PET/MRI in Prostate Cancer Active Surveillance: a Pilot Study
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Recruitment was difficult.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Samuel Joseph Galgano, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R22-145; 300009833 (Other: UAB IRB)
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prostate Cancer (Experimental): 18F-rhPSMA-7.3 PET/MRI in Prostate Cancer Active Surveillance: A Pilot Study
  Interventions: Drug: 18F-rhPSMA-7.3

INTERVENTIONS:
Drug: 18F-rhPSMA-7.3 — 18F-rhPSMA-7.3 PET/MR

SUMMARY:
The purpose of this study is to investigate the usefulness of PET/MRI with an investigational radioactive drug, 18F-rhPSMA-7.3, and MRI contrast in evaluating patients with prostate cancer eligible for active surveillance. This study is for imaging purposes only and is not a treatment study.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-cutaneous malignancy in American men with the majority of men diagnosed with PSA-based screening. As such, many will be found to have low-risk disease when detected early in the disease course. Whole gland radical therapies with primary curative intent are typically invasive and incur a recognized risk of morbidity, particularly in regards to urinary and sexual quality of life measures. For this reason, patients with competing comorbidities or low risk disease have increasingly approached management with active surveillance. The use of active surveillance has increased significantly, particularly in those patients with low-volume, low-grade prostate cancer. For these surveillance protocols, serial PSA biomarker evaluation and periodic repeat prostate biopsies are scheduled to assess for grade or stage progression which may redirect management toward curative treatment options within the window for cure. Since the advent of prostate indication multi-parametric MRI (mpMRI) and its use to target areas of suspicion for biopsy sampling, MRI-TRUS fusion biopsy has been used in the setting of patients with active surveillance to better characterize disease risk stratification for confirmatory biopsy sampling.

Despite the advances mpMRI has offered, its sensitivity for detection of clinically significant prostate cancer is insufficient to replace biopsy at both initial diagnosis and during active surveillance. Additionally, although MRI-TRUS fusion has improved detection of clinically significant cancers, it is known that a fraction of prostate cancers remain occult on mpMRI. Various PSMA radiotracers have been explored as an alternative to mpMRI for the detection of clinically significant prostate cancer. Many of these studies utilize PET/CT, which does not take advantage of the vast superiority of mpMRI over CT and limits their ability to detect clinically significant prostate cancer. However, early studies utilizing PET/MRI (in which the sensitivity of the exam for clinically significant cancer is improved by both the PET and MRI components) have shown promising results. While these studies have explored the role of PSMA-PET/MRI in lesion detection and biopsy guidance, there is little data regarding its use in the setting of active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Men with biopsy-confirmed low risk or favorable intermediate risk prostate cancer who are scheduled to undergo multiparametric prostate MRI and confirmatory biopsy as per institutional active surveillance protocol.

Exclusion Criteria:

* Biopsy-proven prostate cancer not eligible for active surveillance per institutional criteria.
* Current or prior treatment for prostate cancer.
* Suspected prostate cancer without histologic confirmation.
* Inability to undergo 3 Tesla prostate MRI due to claustrophobia and/or MRI- incompatible devices or MR incompatible metal implants.

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of lesions detected in total on the participants' mpMRI exams. | through study completion, average 1 year

SECONDARY OUTCOMES:
Number of lesions detected on the participants' 18F-rhPSMA-7.3 exams. | through study completion, average 1 year

OTHER OUTCOMES:
Number of malignant lesions identified on mpMRI-guided targeted biopsy | through study completion, average 1 year
Number of malignant lesions identified on PET/MRI-guided targeted biopsy | through study completion, average 1 year